CLINICAL TRIAL: NCT05937971
Title: Examination of the Implications of Plantar Sensitivity Training and Aerobic Exercise Training on Balance, Functional Capacity, Gait and Proprioception in Patients With Multiple Sclerosis
Brief Title: Plantar Sensitivity Training and Aerobic Exercise Training in Patients With Multiple Sclerosis (PlaSTAcET Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Arel University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, NAZLI GÜNGÖR, Lecturer, Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PlaSTAcET
Record Dates: First submitted 2023-05-20; First posted 2023-07-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; plantar sensitivity; plantar sensitivity training; aerobic training; clinical trial; balance; gait; functional capacity; proprioception
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plantar sensitivity training group (Experimental): Conventional exercises (with the addition of warm-up and cool-down periods) will be applied to all multiple sclerosis patients participating in the study; In addition, aerobic exercise training will be given. In addition to these exercises, plantar sensory training will be given to the sensory training group. Exercises and plantar sensory training will be given to the participants at intervals of three weeks, with progressively progressive sessions, 2 days a week for 12 weeks. Patients will be evaluated twice, before treatment and at the end of treatment 12 weeks later. Within the scope of the evaluation, balance, functional capacity, gait, proprioception and plantar sensory parameters will be measured in patients.
  Interventions: Other: plantar sensitivity training; Other: aerobic exercise training
- aerobic exercise training group (Active Comparator): Conventional exercises (with the addition of warm-up and cool-down periods) will be applied to all multiple sclerosis patients participating in the study; In addition, aerobic exercise training will be given. In addition to these exercises, plantar sensory training will be given to the sensory training group. Exercises and plantar sensory training will be given to the participants at intervals of three weeks, with progressively progressive sessions, 2 days a week for 12 weeks. Patients will be evaluated twice, before treatment and at the end of treatment 12 weeks later. Within the scope of the evaluation, balance, functional capacity, gait, proprioception and plantar sensory parameters will be measured in patients.
  Interventions: Other: aerobic exercise training

INTERVENTIONS:
Other: plantar sensitivity training — Plantar sensory training protocol:
  Applying a moisturizing cream by washing the feet with warm water and drying them (before coming to the session)
  Dynamic gastro-soleus stretching (20 sec, 5 reps, 2 min)
  Plantar fascia stretch (20 sec, 5 reps, 2 min)
  Picking up sheets with feet (10 reps, 2 min)
  Pushing the small roller under the foot back and forth (10 reps, 2 min)
  Holding the spiny proprioception ball on the plantar surface of the foot while sitting, moving it in anterior-posterior and circular directions (2x2.5 min=5 min)
  Keeping the carpet pieces of different softness and texture on the plantar surface of the foot and moving them in anterior-posterior and circular directions (2x2.5 min=5 min) Soft tissue mobilizations applied to the soles of the feet by the physiotherapist (2 minutes)
  Arms: plantar sensitivity training group
Other: aerobic exercise training — Warm-up exercises; will consist of stretching exercises (20-30 s, 5 repetitions), breathing exercises (6-10 s, 5 repetitions) and range of motion exercises (8-10 s, 5 repetitions) for the whole body. Conventional exercises will include balance (10 s, 5 reps), coordination (5-10 s, 5 reps), stabilization (5-10 s, 5 reps) and strengthening exercises (8-10 s, 5 reps), specific to each patient. Aerobic exercise training was started at 40% of the maximum heart rate on the treadmill and gradually increased at three-week intervals (40% in weeks 1-3, 50% in weeks 4-6, 60% in weeks 7-9, and 70% in weeks 10-12). ) will be progressed. Cool-down exercises will include a gradual lowering of the treadmill speed (3 min) and ankle range of motion exercises. Plantar sensory training begins with a duration of 5 minutes and progresses from a sitting position to a standing position at three-week intervals (1-3 weeks 5 minutes, 4-6 weeks 10 minutes, 7-9 weeks 15 minutes, 10-12 weeks 20 minutes). will be.

SUMMARY:
The aim of this thesis study is to examine whether plantar sensory training given in addition to aerobic exercise training has an additional contribution to balance, functional capacity, walking and proprioception in patients with multiple sclerosis. In this direction, the hypotheses of the study are stated below.

H0 hypothesis: Plantar sensory training given in addition to aerobic exercise training in patients with multiple sclerosis has no additional contribution to balance, functional capacity, walking and proprioception.

H1 hypothesis: Plantar sensory training given in addition to aerobic exercise training in patients with multiple sclerosis has an additional contribution to balance, functional capacity, walking and proprioception.

Conventional exercises (with the addition of warm-up and cool-down periods) will be applied to all multiple sclerosis patients participating in the study; In addition, aerobic exercise training will be given. In addition to these exercises, plantar sensory training will be given to the sensory training group. Exercises and plantar sensory training will be given to the participants at intervals of three weeks, with progressively progressive sessions, 2 days a week for 12 weeks. Patients will be evaluated twice, before treatment and at the end of treatment 12 weeks later. Within the scope of the evaluation, balance, functional capacity, gait, proprioception and plantar sensory parameters will be measured in patients. As a result of the study, it will be examined whether plantar sensory training given in addition to aerobic exercise training in multiple sclerosis patients has an additional contribution to balance, functional capacity, walking and proprioception. There is no study in the literature examining the effects of plantar sensory training and aerobic exercise training on balance, functional capacity, walking and proprioception in patients with multiple sclerosis. In this respect, it is anticipated that the study will contribute to the literature.

DETAILED DESCRIPTION:
The aim of this thesis study is to examine whether plantar sensory training given in addition to aerobic exercise training has an additional contribution to balance, functional capacity, walking and proprioception in patients with multiple sclerosis.

Multiple sclerosis is a chronic progressive neurodegenerative disease that causes damage to neural structures such as myelin sheath, oligodendrocytes, and axons in the central nervous system. In addition to motor, cognitive, cerebellar, visual and brain stem functions, sensory functions are also affected in patients with multiple sclerosis. Loss of deep and superficial senses, dysesthesia and paresthesias can be given as examples of these sensory dysfunctions. It is known that plantar cutaneous sensory information provides important clues in maintaining balance, and disturbances in sensory information for any reason cause postural oscillations. Therefore, it is thought that sensory dysfunction in patients with multiple sclerosis may be related to deficits in maintaining static and dynamic balance. There are limited studies on the positive effects of plantar sensory manipulations on balance in different patient populations.

The decrease in aerobic capacity in patients with multiple sclerosis may affect parameters such as balance, walking, and sensory functions. Due to these effects, activity limitations, decreased walking distance, falls, and injuries related to falling may occur in patients. It has been shown that aerobic exercise training increases functional capacity in patients with multiple sclerosis and deep senses such as proprioception and vibration in different patient groups. In this direction, the aim of the thesis study is to examine whether plantar sensory training given in addition to aerobic exercise training has an additional contribution to balance, functional capacity, walking and proprioception in patients with multiple sclerosis.

There is no study in the literature examining the effects of plantar sensory training and aerobic exercise training on balance, functional capacity, walking and proprioception in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-65
* Being diagnosed with multiple sclerosis according to McDonald's criteria
* EDSS (Expanded Disability Status Scale) score between 3 and 5.5
* Stage 3/4/5 according to functional ambulation classification
* Being able to ambulatory 100 meters independently or with device assistance
* Not having an attack in the last 3 months
* No change in routine treatment for MS (multiple sclerosis) in the past 3 months
* Presence of plantar sensitivity loss (as measured with Semmes-Weinstein monofilaments)

  * having a plantar sensory threshold value higher than 2,83-3.61 for 1st metatarsal head;
  * 2.83-3.61 for 2-3rd metatarsal heads;
  * 2.83-3.61 for 4-5th metatarsal heads;
  * 3.61-4.08 for the lateral and medial heel)(15)
* Decreased functional capacity (6-minute walking test distance F<593±57meters, M<638±44meters) (16)

Exclusion Criteria:

* Being diagnosed with pulmonary, orthopedic or cardiovascular disease
* having diabetic neuropathy
* Having neurological disease other than multiple sclerosis
* Having a diagnosis of root compression, radiculopathy, lumbar disc herniation or complaining of low back pain for the last 3 months(17)
* Using an ankle-foot orthosis (AFO)
* Having cognitive dysfunction (MoCA score <21)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Balance measurement (One-leg standing test(seconds)) | Change from before treatment at 12 weeks of intervention/treatment
  The participant will be asked to stand on one leg while the other's knee is in 90° flexion. The stopwatch will be recorded time in seconds. The test will be terminated if the subject's upper foot touches the ground. Separate measurements are made for both extremities.
Balance measurement (measurement of spatiotemporal parameters of balance (with baropodometry) -Bipedal 30 seconds oscillation amplitude (mm) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to stand on the baropodometry platform surface with both feet. Postural sways will be recorded and it demonstrates the sum of deviations from the center of mass.
Balance measurement (measurement of spatiotemporal parameters of balance (with baropodometry)-Maximum oscillating amplitude (mm) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to stand on the baropodometry platform surface with both feet. Postural sways will be measured and the maximum deviation from the center of mass will be recorded.
Balance measurement (measurement of spatiotemporal parameters of balance (with baropodometry)-Average oscillation rate (mm/s) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to stand on the baropodometry platform surface with both feet. Postural sways will be measured and the average deviation rate from the center of mass will be recorded.
gait measurement (-timed 25-foot walk test) | Change from before treatment at 12 weeks of intervention/treatment
  The T25-FW (timed 25-foot walk test) is a quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the MSFC (Multiple Sclerosis Functional Composite) to be administered at each visit. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
gait measurement(spatiotemporal parameters of gait (with baropodometry) -stride length (mm)) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to walk on the baropodometry platform surface. Stride length will be measured and recorded.
gait measurement spatiotemporal parameters of gait (with baropodometry) -Bilateral maximum pressure (gr/cm2) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to walk on the baropodometry platform surface. The maximum pressure of both feet will be separately measured and recorded.
gait measurement spatiotemporal parameters of gait (with baropodometry) -Bilateral mean pressure (gr/cm2) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to walk on the baropodometry platform surface. The average pressure of both feet will be separately measured and recorded.
gait measurement (spatiotemporal parameters of gait (with baropodometry) -Right-left load distribution (%) (from five different points: 1st metatarsal head, 2nd-3rd metatarsal head, 4th-5th metatarsal head, heel medial, heel lateral) | Change from before treatment at 12 weeks of intervention/treatment
  This measurement will be performed with a baropodometry. The patient is asked to walk on the baropodometry platform surface. Right-left foot load distribution from five different points (1st metatarsal head, 2nd-3rd metatarsal head, 4th-5th metatarsal head, heel medial, heel lateral) will be separately measured and recorded.

SECONDARY OUTCOMES:
functional capacity measurement | Change from before treatment at 12 weeks of intervention/treatment
  6-minute walk test
proprioception measurement (-Ankle position sensation) | Change from before treatment at 12 weeks of intervention/treatment
  Passive motion detection threshold test will be performed with a digital goniometer.
proprioception measurement (-Sensation of ankle kinesthesia) | Change from before treatment at 12 weeks of intervention/treatment
  Joint position reproduction test will be performed with a digital goniometer.

OTHER OUTCOMES:
plantar sensitivity measurement | Change from before treatment at 12 weeks of intervention/treatment
  from 1st metatarsal head, 2nd-3rd. metatarsal head, 4-5. metatarsal head, medial calcaneus, lateral calcaneus points (with Semmes-Weinstein monofilaments)

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Güngör, PT, MSc, Principal Investigator — Istanbul Arel University
Locations (1):
- Istanbul Arel University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Homayuni A, Hosseini Z. Correction: An intervention design for promoting quality of life among patients with multiple sclerosis: a protocol with a planning approach for a mixed methods study. BMC Neurol. 2023 Feb 6;23(1):61. doi: 10.1186/s12883-023-03103-y. No abstract available. PMID 36747125
- [Result] Monaghan AS, Huisinga JM, Peterson DS. The relationship between plantar sensation and muscle onset during automatic postural responses in people with multiple sclerosis and healthy controls. Mult Scler Relat Disord. 2021 Nov;56:103313. doi: 10.1016/j.msard.2021.103313. Epub 2021 Oct 5. PMID 34644600
- [Result] Song Q, Zhang X, Mao M, Sun W, Zhang C, Chen Y, Li L. Relationship of proprioception, cutaneous sensitivity, and muscle strength with the balance control among older adults. J Sport Health Sci. 2021 Sep;10(5):585-593. doi: 10.1016/j.jshs.2021.07.005. Epub 2021 Jul 20. PMID 34293496
- [Result] Peebles AT, Bruetsch AP, Lynch SG, Huisinga JM. Dynamic Balance Is Related to Physiological Impairments in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2018 Oct;99(10):2030-2037. doi: 10.1016/j.apmr.2017.11.010. Epub 2017 Dec 22. PMID 29274726
- [Result] Kalron A, Pasitselsky D, Greenberg-Abrahami M, Achiron A. Do textured insoles affect postural control and spatiotemporal parameters of gait and plantar sensation in people with multiple sclerosis? PM R. 2015 Jan;7(1):17-25. doi: 10.1016/j.pmrj.2014.08.942. Epub 2014 Aug 19. PMID 25153447
- [Result] Naka T, Hayashi T, Sugyo A, Watanabe R, Towatari F, Maeda T. The effects of lower extremity deep sensory impairments on walking capability in patients with incomplete cervical spinal cord injury. J Spinal Cord Med. 2022 Mar;45(2):287-292. doi: 10.1080/10790268.2020.1788879. Epub 2020 Jul 23. PMID 32701408
- [Result] Parsons SL, Mansfield A, Inness EL, Patterson KK. The relationship of plantar cutaneous sensation and standing balance post-stroke. Top Stroke Rehabil. 2016 Oct;23(5):326-32. doi: 10.1080/10749357.2016.1162396. Epub 2016 Mar 31. PMID 27077993
- [Result] Khalifeloo M, Naghdi S, Ansari NN, Akbari M, Jalaie S, Jannat D, Hasson S. A study on the immediate effects of plantar vibration on balance dysfunction in patients with stroke. J Exerc Rehabil. 2018 Apr 26;14(2):259-266. doi: 10.12965/jer.1836044.022. eCollection 2018 Apr. PMID 29740561
- [Result] Chisholm AE, Qaiser T, Williams AMM, Eginyan G, Lam T. Acquisition of a precision walking skill and the impact of proprioceptive deficits in people with motor-incomplete spinal cord injury. J Neurophysiol. 2019 Mar 1;121(3):1078-1084. doi: 10.1152/jn.00432.2018. Epub 2019 Feb 6. PMID 30726165
- [Result] Langeskov-Christensen M, Heine M, Kwakkel G, Dalgas U. Aerobic capacity in persons with multiple sclerosis: a systematic review and meta-analysis. Sports Med. 2015 Jun;45(6):905-23. doi: 10.1007/s40279-015-0307-x. PMID 25739555
- [Result] Van Geel F, Bielen H, Theunissen K, Moumdjian L, Van Nieuwenhoven J, Van Wijmeersch B, Meesen R, Ramari C, Feys P. Clinical manifestation and perceived symptoms of walking-related performance fatigability in persons with multiple sclerosis. Int J Rehabil Res. 2021 Jun 1;44(2):118-125. doi: 10.1097/MRR.0000000000000457. PMID 33534273
- [Result] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Result] Dixit S, Maiya A, Shastry BA. Effects of Aerobic Exercise on Vibration Perception Threshold in Type 2 Diabetic Peripheral Neuropathy Population Using 3-sites Method: Single-blind Randomized Controlled Trial. Altern Ther Health Med. 2019 Mar;25(2):36-41. PMID 30990792
- [Result] Burcal CJ, Wikstrom EA. Plantar Cutaneous Sensitivity With and Without Cognitive Loading in People With Chronic Ankle Instability, Copers, and Uninjured Controls. J Orthop Sports Phys Ther. 2016 Apr;46(4):270-6. doi: 10.2519/jospt.2016.6351. Epub 2016 Jan 26. PMID 26813754
- [Result] Chetta A, Zanini A, Pisi G, Aiello M, Tzani P, Neri M, Olivieri D. Reference values for the 6-min walk test in healthy subjects 20-50 years old. Respir Med. 2006 Sep;100(9):1573-8. doi: 10.1016/j.rmed.2006.01.001. Epub 2006 Feb 7. PMID 16466676
- [Result] Vaitkus A, Sipylaite J. Sensory Perception in Lumbosacral Radiculopathy with Radicular Pain: Feasibility Study of Multimodal Bedside-Suitable Somatosensory Testing. Acta Med Litu. 2021;28(1):97-111. doi: 10.15388/Amed.2021.28.1.18. Epub 2021 Apr 29. PMID 34393632